CLINICAL TRIAL: NCT04719754
Title: Epidemiology and Clinico-investigative Study of Abnormal Vaginal Discharge During Pregnancy
Brief Title: Epidemiology of Abnormal Vaginal Discharge During Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Makarem Hassan, Resident, Assiut University
Other Study IDs: VD-WHH
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Vaginal Infection
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women with abnormal vaginal discharge
  Interventions: Diagnostic Test: Vaginal swab
- Pregnant women without abnormal vaginal discharge
  Interventions: Diagnostic Test: Vaginal swab

INTERVENTIONS:
Diagnostic Test: Vaginal swab — The other vaginal swab will be cultured on blood agar, chocolate agar, MacConkey agar and Sabourauds dextrose agar. The cultures will be incubated at 37ºC for 24-96 h or until the colonies appear.

SUMMARY:
Vaginitis among women of childbearing age is well acknowledged as a public health concern due to its high occurrence. Vulvovaginitis is a disorder of the vulva and/or vagina caused by infection, inflammation, or changes in the flora.

There are many types of infections that affect the vagina, the most common three types of infection: bacterial vaginosis, trichomoniasis, and candidiasis. Bacterial vaginosis is the most common vaginal infection in women of reproductive age causing thin and milky vaginal discharge with a fishy odor. Trichomoniasis causes a frothy, greenish-yellow discharge with a foul smell.

Vaginal Candidiasis is one of the most common fungal infections of the female genital tract and the second most common vaginal infection affecting women of reproductive age (after the bacterial infection worldwide. It affects more than 75% of women at least once in their lifetime, with approximately 50% of them also suffering a single recurrence.

About 75% of patients suffering from candidiasis are asymptomatic, but it may be symptomatic with clinical picture characterized by itching, vaginal pain, vulvar burning sensation, dyspareunia, dysuria and mildly unpleasant odor, erythema and vulvar edema, white-yellowish plaques on the walls of the vagina and cervix and cheesy vaginal discharge. The risk of vulvo-vaginal candidiasis increases by 30% during pregnancy also in pregnancy, the presence of vaginitis is related to abortion, intrauterine infection, fetal growth retardation, premature rupture of membranes, preterm birth, low birth weight, puerperal infection, and other adverse pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* At any gestational age
* Age of patient: 19-40

Exclusion Criteria:

* Women in labor
* Women with current vaginal bleeding
* Women with current preterm rupture of membrane
* Women immunocompromised women
* Women patients who refused to participate in the study

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The prevalence of microorganism in the vaginal discharge during pregnancy. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed K Ibrahim, MD, Study Director — Woman's Health Hospital- Assiut university
Locations (1):
- Woman's Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided